CLINICAL TRIAL: NCT06871696
Title: Genetic of Intellectual Deficiency and Autism Spectrum Disorders
Brief Title: Genetic of Intellectual Deficiency and Autism Spectrum Disorders (RaDiCo-GenIDA)
Acronym: RaDiCo-GenIDA
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C14-35
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Genetic of Intellectual Deficiency; Autism Spectrum Disorder
Keywords: Autism Spectrum; Intellectual Disability; Rare disease; Genetic origin
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Institut National de la Santé et de la Recherche Médicale, France

SUMMARY:
The aim of this observational study is to develop an alternative database model for genetically originated intellectual disabilities. This model will take the form of an online cohort study, where the majority of clinical information will be provided by the families of the patients. Questionnaires developed by professionals but formulated in a way understandable to families will be used to gather this information.

Specifically, this study aims to collect relevant information for personalized medical management. This includes understanding the risks of specific pathological complications and potential iatrogenic effects of symptomatic treatments. The primary goal is to establish groups of individuals with intellectual disabilities and/or autism spectrum disorders (ASD) sharing the same genetic mutation. This approach will provide a better understanding of the natural history of the disease and associated comorbidities.

It is important to note that this project will only focus on patients for whom the identification of the causal mutation or penetrant copy number variation (CNV) has been determined. It excludes individuals for whom the cause of intellectual disability is unknown.

This approach will contribute to a better understanding of the genetic aspects of intellectual disabilities and ASD, while facilitating more targeted and personalized medical care for the affected patients.

ELIGIBILITY:
Inclusion Criteria:

* Be a voluntary adult (aged 18 or older)
* Be a family member (i.e., mother/father) of patients with intellectual disabilities and/or autism spectrum disorders of known genetic origin. This includes monogenic causes as well as recurrent copy number variations (CNVs) such as deletions or duplications. Note: we also allow adult patients to participate directly if they wish and have the capacity to do so.
* Have knowledge of the genetic cause behind intellectual disabilities or autism spectrum disorders. An exception to this rule is possible for patients with a syndrome that includes intellectual disabilities or autism spectrum disorders, and for whom genetic investigation is considered, with the approval of the project's scientific council (which will define the syndromes eligible for this exception).
* Have the intellectual and material capabilities to complete an internet questionnaire.
* Have read the information sheet regarding the study and agreed to the general conditions of participation in the study.

There are no restrictions based on age, gender, or potential comorbidities of the individual themselves.

Exclusion Criteria:

* Patients affected by the presence of intellectual disability and/or an autism spectrum disorder of unknown genetic origin will not be able to participate in the study, except with the exception mentioned in the previous chapter.
* It is requested that only adults enter data. However, the collected data may pertain to a minor (in the case of a parent entering data about their minor child)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The studied population includes all patients (and their relatives*) affected by intellectual disability (ID) and/or autism spectrum disorders (ASD) of known genetic origin, on an international scale.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Description of the clinical and "para-clinical" characteristics of the disease over time in adult and pediatric patients, depending on the type of genetic anomaly associated with the disease. | Day 1, Every 6 months over 5 years

SECONDARY OUTCOMES:
Identification of new information regarding the challenges faced by individuals with Intellectual Disability/Autism Spectrum Disorder (ID/ASD), based on their age (pediatric/adult) and type of anomaly (genetic/environmental factor). | Day 1, Every 6 months over 5 years
Search for associations between certain phenotypic and genotypic/environmental factor characteristics to which individuals have been exposed. | Day 1, Every 6 months over 5 years
Description of the dynamics of exchanges among families (no access to content, description of the number of participating families, frequency of exchanges, etc.) | Day 1, Every 6 months over 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- RaDiCo-GenIDA, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No